CLINICAL TRIAL: NCT01107119
Title: Enabling Elderly Patients to Manage Their Own Lives - A Systematic Management Program for Home Care Services.
Brief Title: Integrated Care Pathways in a Community Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: The Research Council of Norway (Other); St. Olavs Hospital (Other); Nordmøre and Romsdal Hospital Trust (Unknown); City of Trondheim (Unknown); Local authorities of Orkdal (Unknown); Local authorities of Surnadal (Unknown); Local authorities of Sunndal (Unknown); Local authorities of Fræna (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 21528
Record Dates: First submitted 2010-04-18; First posted 2010-04-20 (Estimated); Last update posted 2017-04-20 (Actual); Status verified 2017-04

CONDITIONS: Chronic Illness
Keywords: Frail elderly; Chronic illness; Integrated care model; Clinical pathways; Home care services
MeSH Terms: conditions — Chronic Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Integrated care pathway (Experimental): program for
  1. communication and information flow aimed at collaboration between hospitals, general practitioners and home care services
  2. systematic patient follow-up in home care services by using checklists
  Interventions: Other: integrated care pathway
- usual care (Active Comparator): usual care
  Interventions: Other: usual care

INTERVENTIONS:
Other: integrated care pathway — communication and follow-up program for integrated care
  Arms: Integrated care pathway
Other: usual care
  Arms: usual care

SUMMARY:
The ambition of this study is to raise the quality of care for old and chronically ill patients by establishing a sustainable, systematic prevention and integrated care model for users of home care services.

In this cluster randomized study the intervention will be carried through in five municipalities and three general hospitals. The home care units in every municipality will be randomized to either intervention og control units.

DETAILED DESCRIPTION:
The primary objective of this study is to develop a functional and integrated care model between primary and secondary health care that will meet the needs both in the city and in smaller rural areas.

The secondary objective of this study is to reduce the need of care at primary and secondary level through a a systematic and integrated follow-up by home care nurses and general practitioners to:

* Enable these patients to manage their health needs more efficiently and independently
* Achieve better collaboration within primary care
* Achieve better collaboration between primary- and secondary health care professionals
* Achieve increased satisfaction and confidence with the health care services by the users and their relatives both for included patients and other patients receiving home care services.
* Promote health and prevent unnecessary decline in health
* Strengthen the patients' ability to manage their daily activities.

ELIGIBILITY:
Inclusion Criteria:

* Person 70 years or above being discharged from the general hospital
* Will receive home care services within four weeks after being discharges from the hospital.

Exclusion Criteria:

* Do not agree or are not able to agree to participate
* Is already involved in other research studies affecting the home care services.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 304 (Actual)
Dates: Start 2009-10; Primary Completion 2012-03 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
activities of daily living (ADL) | 6 and 12 months
  Individbasert pleie- og omsorgsstatistikk (IPLOS) scale, and Nottingham Extended ADL Scale
Institutional health care at primary and secondary level | 1 year
  Readmission (30 days)and inpatient hospital stays, number and length of stay (EPJ hospitals) Number and length of stay in municipal nursing homes (EPJ municipals) Days before permanent stay in municipal nursing homes

SECONDARY OUTCOMES:
Achieve better collaboration within primary care and between primary- and secondary health care providers | 1 year
  Extract information on communication from EPJ municipal care and EPJ General practitioners

CONTACTS AND LOCATIONS:
Overall Officials: Anders Grimsmo, md phd, Principal Investigator — Norwegian University of Science and Technology
Locations (7):
- Norway (7):
  - Fræna Municpality, Fræna
  - Molde hospital, Molde
  - Orkdal Municipality, Orkdal
  - Sunndal Municiplaity, Sunndal
  - Surnadal Municipality, Surnadal
  - St Olav's University hospital, Trondheim
  - Trondheim municiplaity, Trondheim

REFERENCES:
- [Background] Rosstad T, Garasen H, Steinsbekk A, Sletvold O, Grimsmo A. Development of a patient-centred care pathway across healthcare providers: a qualitative study. BMC Health Serv Res. 2013 Apr 1;13:121. doi: 10.1186/1472-6963-13-121. PMID 23547654
- [Result] Rosstad T, Garasen H, Steinsbekk A, Haland E, Kristoffersen L, Grimsmo A. Implementing a care pathway for elderly patients, a comparative qualitative process evaluation in primary care. BMC Health Serv Res. 2015 Mar 4;15:86. doi: 10.1186/s12913-015-0751-1. PMID 25888898
- [Result] Rosstad T, Salvesen O, Steinsbekk A, Grimsmo A, Sletvold O, Garasen H. Generic care pathway for elderly patients in need of home care services after discharge from hospital: a cluster randomised controlled trial. BMC Health Serv Res. 2017 Apr 17;17(1):275. doi: 10.1186/s12913-017-2206-3. PMID 28412943